CLINICAL TRIAL: NCT02921087
Title: Connecting Contact Lenses and Digital Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Danielle Iacono, Assistant Clinical Professor, State University of New York College of Optometry
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 923606
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Asthenopia; Contact Lenses; Ocular Accommodation; Convergence, Excess
MeSH Terms: conditions — Asthenopia; Ocular Motility Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test followed by control (Other): Subjects will be randomized in a 1:1 ratio based on a randomization schedule according to sequentially assigned subject numbers to the test daily disposable soft contact lenses at the first visit. Subjects will crossover to the control daily disposable soft contact lenses at the second visit.
  Interventions: Device: Test Daily Disposable Soft Contact Lenses; Device: Control Daily Disposable Soft Contact Lenses
- Control followed by test (Other): Subjects will be randomized in a 1:1 ratio based on a randomization schedule according to sequentially assigned subject numbers to the control daily disposable soft contact lenses at the first visit. Subjects will crossover to the test daily disposable soft contact lenses at the second visit.
  Interventions: Device: Test Daily Disposable Soft Contact Lenses; Device: Control Daily Disposable Soft Contact Lenses

INTERVENTIONS:
Device: Test Daily Disposable Soft Contact Lenses — Worn daily for 7 +/- 2 days
Device: Control Daily Disposable Soft Contact Lenses — Worn daily for 7 +/- 2 days

SUMMARY:
This study seeks to address whether or not different types of daily disposable soft contact lenses may be a beneficial option for patients complaining of eye strain and visual discomfort while using digital devices.

DETAILED DESCRIPTION:
This was a prospective, single site, randomized, double-masked, crossover pilot study. Subjects were randomized to begin with either multifocal or single vision distance contact lenses. The lenses used in this study were the 1-Day Acuvue (AV) Moist spherical single-vision soft contact lenses (SSCL) in the 8.5 base curve and the 1-Day AV Moist Multifocal (MFSCL) in the low ADD (etafilcon A, 58% water content). The preferred viewing distance on digital devices for a similar age group to our study was 63 cm which would require a near ADD of +1.59D. A low addition (ADD) yielding up to +1.25D was selected to provide an intermediate near addition without compromising distance vision as much as would be expected with higher add powers. The multifocal lens utilizes an aspheric center-near design. Subjects wore the lenses on a daily wear, daily disposable schedule. Following one week (± 2 days) of lens wear, subjects were evaluated and the alternate lenses dispensed. Adverse events were collected and assessed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 35 years of age
2. Spectacle prescription of -0.75 to -6.00 D sphere with no more than 0.75 diopters of refractive cylinder
3. Current single-vision soft contact lens wearer
4. Monocular acuity of 20/25 or better in each eye (Snellen)
5. Self-reported minimum of 6 hours a day on digital devices
6. Self-reported complaint of eyestrain on digital devices
7. No ocular pathology and/or history of eye surgery
8. No history of strabismus or strabismus surgery
9. No gas permeable lens wear for at least 3 months
10. Subjects may not be optometrists, opticians or optometry students

Exclusion Criteria:

1. Corneal staining, blepharitis and/or Meibomian Gland Dysfunction (MGD) worse than Grade 2 using the Efron Grading Scale
2. Negative Relative Accommodation (NRA) less than +1.50 D
3. Exophoria at near > 6 prism diopters10
4. Vertical phoria > 1 prism diopter
5. Presence of tropia
6. Response of 3 or higher on question 2b of the Contact Lens Dry Eye Questionnaire- 8 (CLDEQ-8)
7. Unacceptable contact lens fit (i.e. substantially decentered, excessive movement)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Iacono, OD, Principal Investigator — SUNY Optometry
Locations (1):
- SUNY College of Optometry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ember, Sydney. Brands Woo Millennials With a Wink, an Emoji or Whatever It Takes. New York Times 28 September 2015: B1.
- [Background] Rueff, Erin. Contact Lens Induced Dry Eye And Binocular Vision Disorders: A Study Of Similar Symptoms. (2014): Networked Digital Library of Theses & Dissertations. Oct. 2015.
- [Background] Cooper, Jeffrey S., et al. Care of the patient with accommodative and vergence dysfunction. American Optometric Association. USA (1998): 5-10.
- [Background] Rouse MW, Borsting EJ, Mitchell GL, Scheiman M, Cotter SA, Cooper J, Kulp MT, London R, Wensveen J; Convergence Insufficiency Treatment Trial Group. Validity and reliability of the revised convergence insufficiency symptom survey in adults. Ophthalmic Physiol Opt. 2004 Sep;24(5):384-90. doi: 10.1111/j.1475-1313.2004.00202.x. PMID 15315652
- [Background] Chalmers RL, Begley CG, Moody K, Hickson-Curran SB. Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) and opinion of contact lens performance. Optom Vis Sci. 2012 Oct;89(10):1435-42. doi: 10.1097/OPX.0b013e318269c90d. PMID 22960615
- [Background] Jaschinski W. The proximity-fixation-disparity curve and the preferred viewing distance at a visual display as an indicator of near vision fatigue. Optom Vis Sci. 2002 Mar;79(3):158-69. doi: 10.1097/00006324-200203000-00010. PMID 11913842
- [Background] Richdale K, Mitchell GL, Zadnik K. Comparison of multifocal and monovision soft contact lens corrections in patients with low-astigmatic presbyopia. Optom Vis Sci. 2006 May;83(5):266-73. doi: 10.1097/01.opx.0000216098.62165.34. PMID 16699438
- [Background] Fedtke C, Bakaraju RC, Ehrmann K, Chung J, Thomas V, Holden BA. Visual performance of single vision and multifocal contact lenses in non-presbyopic myopic eyes. Cont Lens Anterior Eye. 2016 Feb;39(1):38-46. doi: 10.1016/j.clae.2015.07.005. Epub 2015 Jul 27. PMID 26228543
- [Background] Efron, Nathan. Clinical application of grading scales for contact lens complications. Optician 213.5604 (1997): 26-34.
- [Background] Morgan MW. The clinical aspects of accommodation and convergence. Am J Optom 1944; 21:301-13.
- [Background] Hayes JR, Sheedy JE, Stelmack JA, Heaney CA. Computer use, symptoms, and quality of life. Optom Vis Sci. 2007 Aug;84(8):738-44. doi: 10.1097/OPX.0b013e31812f7546. PMID 17700327

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty five subjects were consented and screened. Twenty three were found to be eligible and randomized. Twenty two completed the study.
Groups:
- Test 1 Week, Followed by Control 1 Week, no Washout: Subjects will be randomized in a 1:1 ratio based on a randomization schedule according to sequentially assigned subject numbers to the test daily disposable soft contact lenses at the first visit. Subjects will crossover to the control daily disposable soft contact lenses at the second visit.
  Test Daily Disposable Soft Contact Lenses: Worn daily for 7 +/- 2 days
  Control Daily Disposable Soft Contact Lenses: Worn daily for 7 +/- 2 days
- Control 1 Week, Followed by Test 1 Week, no Washout: Subjects will be randomized in a 1:1 ratio based on a randomization schedule according to sequentially assigned subject numbers to the control daily disposable soft contact lenses at the first visit. Subjects will crossover to the test daily disposable soft contact lenses at the second visit.
  Test Daily Disposable Soft Contact Lenses: Worn daily for 7 +/- 2 days
  Control Daily Disposable Soft Contact Lenses: Worn daily for 7 +/- 2 days
Period: Overall Study
Arm/Group | Test 1 Week, Followed by Control 1 Week, no Washout | Control 1 Week, Followed by Test 1 Week, no Washout
Started | 12 | 11
Completed | 12 | 10 (One subject dropped out prior to 1 week of lens wear while wearing the control lens (lens 1).)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Followed by Control | Control Followed by Test | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.83 (3.63) | 25.09 (3.48) | 27.04 (3.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 5 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Subjective Symptom Improvement
Description: The primary outcome measure was change in average score on a ten question Visual Comfort Survey using a Visual Analogue Scale (VAS) from baseline to day 7 in multifocal contact lenses and single vision contact lenses. The Visual Analogue Scale ranges from 0-100 (100 being the worst symptoms) for each of the ten questions. The maximum total score is 1000, the minimum total score is 0 (no symptoms).
Time Frame: Baseline and after 1 week of wearing each lens.
Population: Forty five subjects were enrolled into the study. Twenty three eligible subjects were randomized. One subject discontinued early due to discomfort in the first lens assigned. One week data for the primary outcome was available for 22 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Test Arm: Multifocal Soft Contact Lenses: Symptoms after one week of wearing multifocal soft spherical contact lenses.
- Control Arm: Single Vision Spherical Contact Lenses: Symptoms after one week of wearing single vision soft spherical contact lenses.
- Baseline Symptoms: Symptoms at visit one in habitual contact lenses
Arm/Group | Test Arm: Multifocal Soft Contact Lenses | Control Arm: Single Vision Spherical Contact Lenses | Baseline Symptoms
Number analyzed (Participants) | 22 | 22 | 22
score on a scale | 153.9 (124.9) | 100.7 (79.2) | 272.13 (150.19)
Statistical Analysis 1: Comparison: Test Arm: Multifocal Soft Contact Lenses vs Control Arm: Single Vision Spherical Contact Lenses; In order to analyze the 2 x 2 crossover design for the primary outcome (change in overall VAS at day 7) mixed model analysis was utilized, allowing the sequences of each subject to be modeled as repeated measures within PROC Mixed; Test type: Superiority; p = 0.07, Mixed Models Analysis; Least-squares adjusted means were obtained and compared

2. Secondary Outcome: Lens Preference
Description: Based on two alternative forced choice method
Time Frame: 2 weeks
Population: Forty five subjects were enrolled into the study. Twenty three eligible subjects were randomized. One subject discontinued early due to discomfort in the first lens assigned. Data was available for 22 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Preferred Multifocal Lenses: Percentage of subjects who preferred the multifocal (test) lenses
- Preferred Single Vision Lenses: Percentage of subjects who preferred the single vision (control) lenses
Arm/Group | Preferred Multifocal Lenses | Preferred Single Vision Lenses
Number analyzed (Participants) | 22 | 22
Participants | 7 | 15

3. Secondary Outcome: Lag of Accommodation in Study Lenses
Description: Accommodative response was measured by having subjects switch the right lens to a spherical lens in the appropriate power. This was done for all subjects regardless of which lens they were randomized to, to maintain masking. Subjects wore an infrared filter over the right eye for occlusion and to ensure that they were fixating with the left eye (which was still wearing the lens they were randomized to). This filter allowed for measurements to be taken with the WAM-5500 open field autorefractor in front of the right eye. This method assumes a symmetrical accommodative response between eyes. Since accommodative response was measured monocularly, this eliminated any convergent accommodation, but this was consistent between lenses and test distances. Five measurements were taken at each test distance (distance, 40cm and 25cm). The 5 readings obtained were used to calculate mean spherical equivalent value at each test distance and compared to expected accommodative value to determine lag.
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Diopters
Groups:
- Test Arm: Multifocal Soft Contact Lenses: Lag of Accommodation while wearing multifocal soft spherical contact lenses.
- Control Arm: Single Vision Spherical Contact Lenses: Lag of Accommodation while wearing single vision soft spherical contact lenses.
Arm/Group | Test Arm: Multifocal Soft Contact Lenses | Control Arm: Single Vision Spherical Contact Lenses
Number analyzed (Participants) | 22 | 22
Diopters
  Lag at 25 cm | 1.52 (0.47) | 1.23 (0.57)
  Lag at 40 cm | 1.06 (0.60) | 0.75 (0.45)
  Lag at Distance | 0.00 (0.43) | 0.22 (0.44)
Statistical Analysis 1: Comparison: Test Arm: Multifocal Soft Contact Lenses vs Control Arm: Single Vision Spherical Contact Lenses; In order to analyze the 2 x 2 crossover design for accommodative response mixed model analysis was utilized, allowing the sequences of each subject to be modeled as repeated measures within PROC Mixed; Test type: Superiority; p = 0.01, Mixed Models Analysis; Least-squares adjusted means were obtained and compared

4. Secondary Outcome: Convergence Insufficiency Symptom Survey (CISS)
Description: Difference in CISS score after one week of multifocal contact lens use vs single vision contact lens use. Minimum score (least symptoms)= 0. Maximum score (worst symptoms) = 60.
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Arm: Multifocal Soft Contact Lenses | Control Arm: Single Vision Spherical Contact Lenses
Number analyzed (Participants) | 22 | 22
score on a scale | 11.2 (6.8) | 10.8 (5.6)
Statistical Analysis 1: Comparison: Test Arm: Multifocal Soft Contact Lenses vs Control Arm: Single Vision Spherical Contact Lenses; In order to analyze the 2 x 2 crossover design for the change in CISS, mixed model analysis was utilized, allowing the sequences of each subject to be modeled as repeated measures within PROC Mixed; Test type: Superiority; p = 0.77, Mixed Models Analysis; Least-squares adjusted means were obtained and compared

5. Secondary Outcome: Contact Lens Dry Eye Questionnaire- 8 Survey (CLDEQ-8)
Description: CLDEQ-8 score after one week of multifocal contact lenses vs single vision contact lenses. Minimum value (least symptoms) = 0. Maximum Score= 37 (worst symptoms).
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Arm: Multifocal Soft Contact Lenses | Control Arm: Single Vision Spherical Contact Lenses
Number analyzed (Participants) | 22 | 22
score on a scale | 11.7 (6.4) | 11.0 (4.7)
Statistical Analysis 1: Comparison: Test Arm: Multifocal Soft Contact Lenses vs Control Arm: Single Vision Spherical Contact Lenses; In order to analyze the 2 x 2 crossover design for the CLDEQ-8, mixed model analysis was utilized, allowing the sequences of each subject to be modeled as repeated measures within PROC Mixed; Test type: Superiority; p = 0.69, Mixed Models Analysis; Least-squares adjusted means were obtained and compared

6. Secondary Outcome: Near Phoria at 40cm in Multifocal Contact Lens vs Single Vision Contact Lens
Description: Measured via Modified Thorington
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Prism Diopters of Exophoria
Groups:
- Test Arm: Multifocal Soft Contact Lenses: Near Phoria while wearing multifocal soft spherical contact lenses.
- Control Arm: Single Vision Spherical Contact Lenses: Near Phoria while wearing single vision soft spherical contact lenses.
Arm/Group | Test Arm: Multifocal Soft Contact Lenses | Control Arm: Single Vision Spherical Contact Lenses
Number analyzed (Participants) | 22 | 22
Prism Diopters of Exophoria | 2.3 (3.8) | 2.0 (4.5)
Statistical Analysis 1: Comparison: Test Arm: Multifocal Soft Contact Lenses vs Control Arm: Single Vision Spherical Contact Lenses; In order to analyze the 2 x 2 crossover design for phoria, mixed model analysis was utilized, allowing the sequences of each subject to be modeled as repeated measures within PROC Mixed; Test type: Superiority; p = 0.87, Mixed Models Analysis; Least-squares adjusted means were obtained and compared

7. Post Hoc Outcome: Participants Stratified by Subjects' Near Phoria With Single Vision Lenses
Time Frame: 1 week
Population: Phoria at near as measured through the single vision spherical contact lenses
Measure: Count of Participants; unit: Participants
Groups:
- Phoria in Single Vision Spherical Contact Lenses: Phoria at near as measured through the single vision spherical contact lenses
Arm/Group | Phoria in Single Vision Spherical Contact Lenses
Number analyzed (Participants) | 22
Participants
  Esophoria at Near | 5
  Exophoria/ Orthophoria at Near | 17

8. Post Hoc Outcome: Phoria and Lens Preference
Description: Subjects' phoria at near with single vision lenses was classified as esophoric or exophoric. Lens preference was compared (multifocal vs single vision lenses) between the subjects who were esophoric at near vs the subjects who were exophoric/orthophoric at near.
Time Frame: 1 week
Population: Forty five subjects were enrolled into the study. Twenty three eligible subjects were randomized. One subject discontinued early due to discomfort in the first lens assigned. Of the 22 completed subjects, 5 had an esophoria at near. 17 were exophoric or orthophoric at near.
Measure: Count of Participants; unit: Participants
Groups:
- Esophoric at Near: Subjects who are esophoric at near with single vision contact lenses
- Exophoric or Orthophoria at Near: Subjects who were exophoric or orthophoric at near in single vision contact lenses
Arm/Group | Esophoric at Near | Exophoric or Orthophoria at Near
Number analyzed (Participants) | 5 | 17
Participants
  Preferred Multifocal Contact Lenses | 5 | 2
  Preferred Single Vision Contact Lenses | 0 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study, which lasted for approximately 2 weeks per subject.
Groups:
- Multifocal Contact Lenses: Adverse Events while wearing Multifocal Contact Lenses
- Single Vision Contact Lenses: Adverse Events while wearing Single Vision Contact Lenses
Arm/Group | Multifocal Contact Lenses | Single Vision Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 2/22 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multifocal Contact Lenses (N=22) | Single Vision Contact Lenses (N=23)
Conjunctival Hyperemia (Eye disorders) | 0 (0) | 1 (2) — Occurred after lens removal
Cold Like Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subcojnunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02921087/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT02921087/SAP_001.pdf